CLINICAL TRIAL: NCT06053398
Title: Vasopressor Outcomes in Spine Surgery
Acronym: V-SPINE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Siddharth Dave, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0326
Record Dates: First submitted 2023-08-31; First posted 2023-09-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypotension
Keywords: Vasopressor; Phenylephrine; Norepinephrine; Spine Surgery; General Anesthesia
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenylephrine (Active Comparator): Patients receiving phenylephrine for intraoperative hypotension
  Interventions: Drug: Phenylephrine
- Norepinephrine (Active Comparator): Patients receiving norepinephrine for intraoperative hypotension
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — Intraoperative phenylephrine infusion Phenylephrine infusion to be titrated as needed to target a mean arterial pressure (MAP) > 65 mm Hg.
  Arms: Phenylephrine
Drug: Norepinephrine — Intraoperative norepinephrine infusion Norepinephrine infusion to be titrated as needed to target a MAP > 65 mm Hg.
  Arms: Norepinephrine

SUMMARY:
This is a prospective, randomized control trial comparing norepinephrine versus phenylephrine for vasopressor support in patients undergoing elective spinal fusion surgery.

DETAILED DESCRIPTION:
There is limited evidence on the difference in postoperative outcomes between the choices of vasopressors used to treat intraoperative hypotension (IOH) in patients undergoing non-cardiac surgery under general anesthesia. A recent pilot feasibility trial comparing norepinephrine and phenylephrine for first-line intravenous infusion of vasopressor during general anesthesia and major non-cardiac surgery was unable to show any difference in postoperative outcomes. Although the study demonstrated safety and feasibility, it was not powered to detect differences in postoperative outcomes. The impact of vasopressors on postoperative outcomes in patients undergoing complex spinal surgery in the prone position is even scarcer. While it has been demonstrated that the use of intra-operative vasopressor infusion is safe and well tolerated, without any adverse renal outcomes, it is unclear if the choice of vasopressor makes any difference. While animal studies have shown that norepinephrine may provide greater spinal cord protection than phenylephrine, clinical studies in humans are lacking. We aim to fill this gap in knowledge by carrying out a prospective, randomized control trial to evaluate differential outcomes related to the choice of norepinephrine versus phenylephrine as the preferential vasopressor in patients undergoing elective spinal fusion surgery in the prone position.

ELIGIBILITY:
Inclusion Criteria:

-Patients > 18 years undergoing elective, prone, spinal fusion surgery

Exclusion Criteria:

* Age < 18 years
* Emergency surgery
* Outpatient surgery
* Pregnancy
* End-stage renal disease requiring dialysis
* Diagnosed myocardial ischemia and/or cardiac revascularization within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Vasopressor requirement | During inpatient admission
  Total intraoperative vasopressor requirement

SECONDARY OUTCOMES:
Postoperative acute kidney injury | During inpatient admission
  Kidney Disease Improving Global Outcomes (KDIGO) criteria
  Acute Kidney Injury (AKI) is defined as any of the following:
  1. Increase in serum creatinine (sCr) ≥0.3 mg/dL (≥26.5 μmol/L) within 48 hours; or
  2. Increase in sCr ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  3. Urine volume <0.5 mL/kg/h for 6 hours
Intraoperative transfusion requirement | During inpatient admission
Postoperative vasopressor requirement | During inpatient admission
Length of ICU stay | During inpatient admission
Length of hospital stay | From admission to discharge (up to 100 weeks)
30-day readmission | 30-days post-discharge
Postoperative Myocardial Injury | During inpatient admission
  Troponin elevation (ng/L)
Postoperative Lactate Elevation | During inpatient admission
  Lactate (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Dave, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Clements University Hospital at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No